CLINICAL TRIAL: NCT05845983
Title: Lactobacillus Acidophilus Improves the Prognosis (Cognitive Function) of Patients With Ischemic Cerebrovascular Disease After Surgery: a Multicenter, Prospective, Three-blind, Placebo-randomized Controlled Study
Brief Title: LA Improves the Prognosis of Patients With ICVD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huaqiu Zhang (Other)
Responsible Party: Sponsor-Investigator, Huaqiu Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ-IRB20230304
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Ischemia; Cerebrovascular Ischemia; Cognitive Impairment
MeSH Terms: conditions — Ischemia; Cerebral Infarction; Cognitive Dysfunction | interventions — Lacteol; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The patient received conventional treatment and Maltodextrin treatment (placebo) for three months after surgery.
  Interventions: Dietary Supplement: Maltodextrin
- LA treatment group (Experimental): The patient received conventional treatment and Lactobacillus acidophilus treatment for three months after surgery.
  Interventions: Dietary Supplement: Lactobacillus acidophilus

INTERVENTIONS:
Dietary Supplement: Lactobacillus acidophilus — Lactobacillus acidophilus solid drink (pure bacteria, food grade, JYLA-191, Shandong Zhongke Jia-yi Biological Engineering Co., LTD.), 3g (containing 2*10^10CFU), twice a day, once in the morning and once in the evening, 1 bag each time, by drinking water, direct oral intake, 1 month/course, continuous use for three courses.
  Arms: LA treatment group
Dietary Supplement: Maltodextrin — Maltodextrin solid drink (food grade, MD20, Shandong Zhongke Jia-yi Biological Engineering Co., LTD.), 3g, twice a day, once in the morning and once in the evening, 1 bag each time, by drinking water, direct oral intake, 1 month/course, continuous use for three courses.
  Arms: Control group

SUMMARY:
Ischemic cerebrovascular disease will cause serious harm to the life and safety of patients, and the treatment prognosis is poor. Numerous clinical trials have demonstrated that probiotics can improve cognitive function in people under multimodal. We have previously found that Lactobacillus acidophilus administration could improve cognitive impairment in MCAO and BCAS mice. Therefore, Based on the above research background and the basis of previous studies, we believe that the administration of Lactobacillus acidophilus solid drink (pure Lactobacillus acidophilus strain) can improve the cognitive function of patients with cerebral ischemia through the "brain-gut axis".

DETAILED DESCRIPTION:
Ischemic cerebrovascular disease, as a common form of stroke, is one of the main causes of global morbidity and mortality. The mortality rate of this disease is relatively high, and the treatment prognosis is poor, which will cause serious harm to the life and safety of patients. The optimal treatment for ischemic cerebrovascular disease is still unclear, and the effects of different treatments are still controversial. Therefore, it is of great clinical significance to explore a safe and simple adjuvant treatment method to help patients recover their nervous system function faster and better.

At present, numerous clinical trials have demonstrated that probiotics can improve cognitive function in people under multimodal. Adding intestinal probiotics can improve the intestinal flora distribution, and significantly improve cognitive function in elderly patients with mild cognitive impairment and prevention of brain atrophy. Lactobacillus acidophilus is rich in short chain fatty acids (SCFA). Clinical studies have shown that SCFA levels are negatively correlated with the severity and prognosis of ischemic stroke. Numerous studies have demonstrated that the intestinal supply short chain fatty acids can improve cognitive function, in the middle cerebral artery occlusion (MCAO) induced by acute cerebral ischemia model, rich in the intestines of SCFA can cure acute cerebral ischemia in mice induced by nerve injury. More importantly, in mice with acute cerebral ischemia induced by middle cerebral artery occlusion (MCAO) and chronic cerebral ischemia caused by bilateral common carotid artery stenosis (BCAS), we have previously found that mice have cognitive impairment, accompanied by intestinal flora dysregulation.

Lactobacillus acidophilus administration has a significant effect on improving cognitive function. Based on the above research background and the basis of previous studies, the researchers believe that the administration of Lactobacillus acidophilus solid drink (pure Lactobacillus acidophilus strain) can improve the cognitive function of patients with cerebral ischemia through the "brain-gut axis", and increase the reliability and scope of revascularization, and ultimately improve the prognosis of patients with ischemic cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Between 35 and 65 years old;
2. Han nationality;
3. Diagnosed as ischemic cerebrovascular disease with mild to moderate symptoms;
4. Can communicate normally, complete neuropsychological tests independently, and sign informed consent;
5. No previous surgical history;
6. No contraindications such as PET, MRI and DSA;
7. No history of stroke identified by imaging;
8. No family history of other chronic diseases, cancer, mental illness or dementia;
9. Improved Rankin scale score ≤2;
10. Ischemic symptoms appeared in the carotid area ≤3 months before the visit;
11. In line with the surgical treatment of ischemic cerebrovascular disease;

Exclusion Criteria:

1. previous dementia;
2. hearing or visual impairment;
3. Drugs that may or are known to influence cognitive abuse;
4. alcohol addiction;
5. Diagnosis of depression, schizophrenia and other psychiatric diseases;
6. MRI showed severe cerebral infarction;
7. Those allergic to Lactobacillus acidophilus;
8. Baseline CT showed intracranial hemorrhage;
9. ischemic onset accompanied by epilepsy;
10. illiteracy;
11. pregnancy or breastfeeding;
12. any serious medical condition that may interact with treatment;

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2023-05-04 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini-mental State Examination (MMSE, 0-30) scale | Three months.
  Higher scale scores mean better cognitive function.
Montreal Cognitive Assessment (MoCA, 0-30) scale | Three months.
  Higher scale scores mean better cognitive function.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang Y, Zhang X, Yu C, Liu Y, Kang H, Liu Y, Ni Y, Xia Y, Jiang Z, Chen J, Zhao K, Han L, Zou X, Wang J, Lei T, Gan C, Zhang H. Lactobacillus acidophilus promotes cognitive function recovery via regulating microglial peroxisomal function in cerebral ischemia. Cell Host Microbe. 2025 Sep 10;33(9):1484-1501.e12. doi: 10.1016/j.chom.2025.07.018. Epub 2025 Aug 13. PMID 40812303